CLINICAL TRIAL: NCT00067067
Title: Circulating Endothelial Progenitor Cells in Gliomas
Brief Title: Investigating Endothelial Precursor Cells (EPCs)
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030269; 03-N-0269
Record Dates: First submitted 2003-08-08; First posted 2003-08-11 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-10

CONDITIONS: Central Nervous System
Keywords: Glioma; Brain Tumor; Endothelial Progenitor Cells
MeSH Terms: conditions — Glioma; Brain Neoplasms

SUMMARY:
Recent studies suggest that cells in the bone marrow-endothelial precursor cells (EPCs)-can provide a blood supply to cancerous tumors.

The purpose of this study is to collect brain tumor and blood samples to look for these EPCs in the samples and analyze the growth signals that may help blood vessels to grow in tumors. Researchers will study the following in the samples: 1) the number of blood vessels in the tumor; 2) the levels of growth factors in the tumor and blood; 3) the levels of circulating EPCs in the blood; and 4) the changes in the genes and proteins in the blood and tumor that influence growth factor levels.

Participants will be 18 years of age or older and have evidence of a brain tumor that requires surgery. From this surgery they will donate blood and tumor samples. Participants will have follow-up visits 4 to 8 weeks after surgery, then at 3-month intervals for two-and-one-half years, then at 6-month intervals thereafter. At these visits, participants will undergo a physical exam, a brain scan, and blood work.

DETAILED DESCRIPTION:
Angiogenesis, or the development of new blood vessels, appears to be one of the keys to tumor survival. Areas of new blood vessel growth, or neovascularization, such as with trauma or tissue ischemia, appear to release factors that stimulate production of endothelial cells from progenitor stem cells located in the bone marrow. Endothelial cells for the inside lining of blood vessels are important in the formation of viable and functional blood vessel conduits. Recent work suggests that tumors-including primary brain tumors-secrete many of the same stimulatory growth factors as normally incite endothelial cells to be produced and turned out into the circulation. Initial evidence suggests that these circulating endothelial progenitor cells (EPCs) play a role in the impressive neovascularization seen with tumors. In this study, we wish to investigate the interaction of gliomas and EPCs to elucidate a potential role for EPCs in tumor formation, response to therapy, progression, and overall survival, as well, to identify potential new targets for anti-tumor and/or anti-angiogenic therapies using genomic and proteomic techniques.

Patients suspected of having, or with prior biopsy proof of, a WHO grade II-IV central nervous system (CNS) glial tumor(s) seen in the Surgical Neurology Branch, NINDS, will be considered for entry into this study. Tissue samples of tumor resected as part of standard care will be collected at surgery and preserved for research. Blood samples will also be collected. Blood will also be collected from anonymous normal volunteers who donate blood at the NIH Blood Bank; these anonymous donors will serve as controls.

ELIGIBILITY:
Inclusion Criteria

1. Radiographic evidence of a primary glial neoplasm of the CNS (WHO grade II-IV) or any patient with a known primary neoplasm of the CNS.
2. Medically indicated (diagnostic and/or therapeutic) tumor resection.
3. Informed consent from patient, age 18 or older to 75 years of age.
4. No racial or ethnic group or gender is excluded.

Exclusion Criteria

1. Inability to provide informed consent prior to surgery.
2. Medical conditions that cannot be corrected prior to surgery that would be standard contraindications for neurosurgery.
3. Pregnant Women: Women of child-bearing age will be tested before surgery for pregnancy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84
Dates: Start 2003-08; Study Completion 2004-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Louis DN, Pomeroy SL, Cairncross JG. Focus on central nervous system neoplasia. Cancer Cell. 2002 Mar;1(2):125-8. doi: 10.1016/s1535-6108(02)00040-5. No abstract available. PMID 12086870
- [Background] Maher EA, Furnari FB, Bachoo RM, Rowitch DH, Louis DN, Cavenee WK, DePinho RA. Malignant glioma: genetics and biology of a grave matter. Genes Dev. 2001 Jun 1;15(11):1311-33. doi: 10.1101/gad.891601. No abstract available. PMID 11390353
- [Background] Asahara T, Murohara T, Sullivan A, Silver M, van der Zee R, Li T, Witzenbichler B, Schatteman G, Isner JM. Isolation of putative progenitor endothelial cells for angiogenesis. Science. 1997 Feb 14;275(5302):964-7. doi: 10.1126/science.275.5302.964. PMID 9020076